CLINICAL TRIAL: NCT04175795
Title: Effectiveness of a Personalized Health Profile on Specificity of Self-Management Goals Among People Living With HIV in Canada: A Blinded Pragmatic Randomized Controlled Trial
Brief Title: Effectiveness of a Personalized Health Profile on Specificity of Self-Management Goals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Principal Investigator, Nancy Mayo, James mcGill Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ABHN_Goals
Record Dates: First submitted 2019-11-19; First posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Chronic Disease; Goals
Keywords: Goal-setting; Goal specificity; Chronic conditions; Health outcome profile
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: A blinded, stratified, randomized, controlled trial design will be used to assess the impact of the personalized health profile on number and specificity of person-defined self-management goals. All participants in the BHN2 cohort will be randomized into one of two groups, the intervention and control group. Participants will be stratified based on gender and number of visits (i.e., whether 1 visit or 2 visits) they had or will attend. Randomization will be done through the computer by the study statistician using randomization.com. All participants enrolled in the parent trial (BHN1) have a numerical ID. The new participants who will be recruited for the BHN2 will be enumerated and then the numbers will be randomized.
Who Masked: Investigator, Outcomes Assessor
Masking Description: For this study, it will not be possible to blind the participants as the intervention is their personalized health profile. To avoid bias in measure, those collecting and analyzing the data will be kept blind to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dashboard group (Experimental): The intervention group will receive their personal profile via this e-mail along with instructions on goal-setting and tips to improve brain health.
  Interventions: Behavioral: My Personal Brain Health Dashboard
- No Dashboard group (No Intervention): The control group will receive only the goal-setting instructions and tips.

INTERVENTIONS:
Behavioral: My Personal Brain Health Dashboard — The intervention of this study is grounded in the knowledge-to-action framework (Graham et al., 2006) and consists of providing feedback by sending participants their personalized health outcome profiles. As mentioned above, the context of our study is the BHN cohort. For all participants enrolled in the parent study, data on wide spectrum of health outcomes have been gathered. As part of the knowledge translation plan, a personalized profile of specific modifiable health outcomes called as "My Personalized Brain Health Profile" has been created for each participant (Appendix B). The profile covers information on brain health outcomes, health and quality of life ratings, and lifestyle factors.
  Arms: Dashboard group

SUMMARY:
With a growing number of people living with chronic diseases, the need to empower people for self-management is rising. A key element in self-management is goal setting but the extent to which meaningful actionable goals (i.e., SMART) can be set without direction from the health care team is not known. Providing people with specific feedback on actionable health outcomes may stimulate the setting of specific goals. To this end, a health outcome profile was computer generated from the existing outcome measures, at first and last recorded visits, of each person enrolled in the Positive Brain Health Now (+BHN) cohort from 5 sites in Canada. This profile will be tested with BHN participants who agreed to enrolled in sub-studies. The main outcome will be the extent to which goals are SMART by using specific words and actionable verbs. A measurement framework and an initial lexical (i.e., collection of vocabularies) has been developed for the goal evaluation. Using text mining techniques (i.e., tokenizing and pos-tagging), the specific components of each goal will be extracted and compared to the lexical using regular expression algorithms. The result will provide information on the specificity of participants' defined goals.

DETAILED DESCRIPTION:
Introduction: With a growing number of people living with chronic diseases, the need to empower people to self-manage their condition is rising. A key element in self-management is goal setting, however, it is not known to what extent people living with chronic conditions are capable of setting their own actionable health-related goals. One possible strategy to improve goal-setting skills is to provide people with specific information about their health profile to stimulate the setting of specific goals. This study contributes to the understanding of the specificity of patient-formulated self-management goals by testing the effectiveness of providing feedback using a personalized health outcome profile.

Objective: To estimate among people living with HIV, to what extent providing feedback on their health outcomes, compared to no feedback, will affect number and specificity of person-defined self-management goals.

Design: A blinded, stratified, randomized controlled trial design will be conducted targeting all participants in the BHN2 (Action for Positive Brain Health Now) cohort in Canada.

Methods: A personalized health outcome profile has been produced for each person enrolled in the BHN1 cohort (Positive Brain Health Now) at cohort entry and at the last recorded visit. The same profile will be developed for the participants who will enroll in the BHN2 as they go through their visits. The profile covers information on brain health outcomes, health and quality of life ratings, and lifestyle factors. Participants from the BHN1 who agreed to enroll in the BHN2 as well as the new participants will be contacted. The intervention group will receive their personal profile along with instructions on goal-setting and tips to improve brain health; the control group will receive only the goal-setting instructions and tips. Over 800 members of the BHN cohort have sufficient data to generate the profile and will be recruited into the study. Persons will be instructed to enter their goals on a specialized web-based goal setting platform within 2 weeks of receiving their profile. At the close of the two-week period, the control group will receive their profile. Text mining techniques will be used to extract information from the person-defined goals and the specificity of the goal will be scored based on word matches to a developed goal-setting lexical.

Expected Results: The expectation is that the intervention group will set more goals and have more words matching the developed lexical than the control group. The total number of words per person-goal will be calculated for each group and Poisson regression will be used to estimate the rate ratio and 95% confidence intervals and compare rate ratios between men and women using an interaction term.

Conclusion: The effect of providing outcome feedback on setting effective self-management goals will be tested in this study. The results will provide a thorough understanding of the quality of person-defined goals using text mining. Moreover, this study provides evidence necessary for future studies using text mining as an inexpensive and timely way for evaluation of textual information.

ELIGIBILITY:
This study is a sub-study under the BHN trial. Eligibility criteria for the main BHN trial includes:

Inclusion Criteria:

* adults age ≥ 35 who have been diagnosed as HIV positive for at least one year, - able to communicate adequately in French or English,
* and able to give an informed consent

Exclusion Criteria:

* dementia,
* life expectancy of <3 years or other,
* non-HIV-related neurological disorder,
* known active central nervous system opportunistic infection or hepatitis C requiring Interferon treatment,
* known Psychotic disorder,
* current (within the past 12 months) substance dependence or abuse.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Goal specificity | "4 weeks" in total for each participant
  The main outcome in this study is the specificity of self-management goals. For goal specificity, text mining techniques will be used. This outcome will be reported as a time-independent discrete variable - number of specific words (matched to a developed lexical) per person-goals.
Number of self-management goals | "4 weeks" in total for each participant
  For this outcome number of goals per person as well as total number of goals per group will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No